CLINICAL TRIAL: NCT03901742
Title: Effect of the Administration of an Enteral Milk Supplemented With Proteins to Infants Admitted in a Pediatric Intensive Care Unit
Brief Title: Usefulness of Protein-enriched Infant Formula in Pediatric Intensive Care.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Maternal, Neonatal and Child Health Research Network (Other); European Regional Development Fund (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FIBHGM-ECNC011-2010
Record Dates: First submitted 2019-03-25; First posted 2019-04-03 (Actual); Last update posted 2019-08-22 (Actual); Status verified 2019-08

CONDITIONS: Protein-Energy Malnutrition
Keywords: Children; Intensive Care; Nutrition; Enteral feeding; Protein intake; Protein balance.; Lean Body Mass
MeSH Terms: conditions — Protein-Energy Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard Enteral Nutrition (Active Comparator): Standard Enteral Nutrition: cow's milk based infant formula (Nidina, Nestlé, Barcelona, Spain).
  Interventions: Other: Standard Enteral Nutrition
- Protein-enriched nutrition (Active Comparator): Protein-enriched Enteral Nutrition: polymeric infant formula (Infatrini; Nutricia, Madrid, Spain)
  Interventions: Other: Protein-enriched nutrition
- High Protein-enriched Nutrition (Active Comparator): High Protein-enriched Enteral Nutrition: polymeric infant formula (Infatrini; Nutricia, Madrid, Spain) supplemented with 2.6 g of protein/100 mL of formula. The source of the protein supplement would be a nonhydrolyzed protein cow's milk-based formula (Resource Protein Instant; Nestlé, Barcelona, Spain). Final composition 5.1 g/100 mL.
  Interventions: Dietary Supplement: High Protein-enriched Nutrition

INTERVENTIONS:
Other: Protein-enriched nutrition — Protein-enriched enteral nutrition with a polymeric infant formula
  Arms: Protein-enriched nutrition
Dietary Supplement: High Protein-enriched Nutrition — High protein-enriched enteral nutrition with a polymeric infant formula plus a protein supplement
  Arms: High Protein-enriched Nutrition
Other: Standard Enteral Nutrition — Cow's milk based infant formula.
  Arms: Standard Enteral Nutrition

SUMMARY:
A multicenter prospective randomized controlled trial (RCT) will be performed in three hospitals. Patients meeting inclusion criteria will be randomly allocated to one of three enteral feeding formula with different protein content. Blood and urine test, nitrogen balance assessment and energy expenditure testing by indirect calorimetry will be performed at the beginning of nutrition regimen and at 24 hours, 72 hours and 5-7 days after initiation. The sample size for this trial is estimated as 90 participants, with approximately 30 participants in each group. The data analysis will be by intention to treat. This RCT will provide new data about the amount of protein needed to improve levels of serum protein and nitrogen balance, surrogate of protein balance, in critically ill infants receiving enteral nutrition.

DETAILED DESCRIPTION:
Background Protein-caloric malnutrition, with an incidence of 15-20 %, is the most important type of malnutrition in Pediatric Intensive Care Units (PICU). It is associated to poor outcomes in critically ill children: malnourished patients present an increased physiologic instability and quantity of care, with higher duration of mechanic ventilation and length of stay and increased mortality.

Current recommendations about protein prescription in critically ill children are fundamentally based on expert opinions, since studies on protein supplementation are scarce, with small sample sizes and heterogeneous patient populations, doses of protein and route of administration.

Study design Once an eligible patient is admitted to PICU, written informed consent will be requested from parents or legal representative of the child by the physician responsible of the patient. They will be made aware that participation is voluntary, and they will be allowed to refuse further participation in the trial whenever they want.

After enrolment, the patient will be allocated randomly, in order of recruitment, into one of the three 3 diet groups using a randomized data table generated with Epidat 3.1 software. A copy of the randomization list will be securely stored in an envelope located at PICU working area desk drawer, which will be opened after the patient enrolment on the study. Physicians, care givers and investigators will know the allocation prior to the start of enteral feeding.

All patients will receive exclusively enteral nutrition via nasogastric o transpyloric tube.

Since this is an open-label trial, the assigned diet will be written down on the medical prescription of each patient and will be prepared by the PICU staff at the own unit, using for it the branded bottles where the different formula are commercialized.

Continuous enteral nutrition will be initiated within the first 24 hours of PICU admission, by transpyloric or nasogastric tube, at a rate of 0.5-1 ml/kg/hour, with increases of 0.5-1 ml/kg every 3-4 hours, if well tolerated, to reach a caloric intake of 60-65 kcal/kg/day, or as needed based on resting energy expenditure measured by indirect calorimetry Demographic data will be recorded at inclusion: gender, age, weight, height, and diagnosis on admission. The risk of mortality at admission will be calculated using pediatric scales: Pediatric Index of Mortality 2 (PIM2), Pediatric Risk of Mortality (PRISM), and Pediatric Logistic Organ Dysfunction (PELOD).

Blood concentrations of urea, creatinine, total proteins, albumin, prealbumin, transferrin, retinol-binding protein (RBP) levels, urinary concentration of urea in 24-hours or isolated urine sample, and energy expenditure, oxygen consumption (VO2) and carbon dioxide production (VCO2) by indirect calorimetry (Datex S5 monitor, E-COVX; General Electrics Healthcare/Datex-Ohmeda, Helsinki, Finland) will be measured at admission and at days 1, 3 and 5-7 after initiation of enteral feeding. Air leaks will be measured using the mechanical ventilator. Calorimetry-derived data will be collected only in patients with tracheal intubation, when air leakage is <10 %, fraction of inspired oxygen (FiO2) less than 80 %, absence of inhaled nitric oxide, sevoflurane or heliox, or connection to extracorporeal membrane oxygenation (ECMO). The collection of indirect calorimetry data will be done over 30 to 120 minutes.

Nitrogen Balance (NB) will be calculated as: nitrogen intake minus total nitrogen losses. Total nitrogen losses will include total urinary nitrogen and fecal/miscellaneous losses estimated according to the World Health Organization recommendations.

Other blood biochemical parameters as glucose, cholesterol, triglycerides, ions and blood gas will also be recorded.

Total daily enteral energy and protein delivery, intravenous albumin infused, and other treatments such as vasoactive drugs, neuromuscular blockers, sedatives and analgesic drugs, diuretics and steroids would be registered.

Protein-enriched diet safety Enteral complications (constipation, diarrhoea, abdominal distension, gastric residue), serum urea and total protein levels, as well as any unexpected adverse event occurring during the trial will be recorded to evaluate the safety of the protein-enriched diet.

Statistical analysis As there are not previous studies reporting expected standard deviations, the standardized difference of means for computing the optimal minimum number of patients to include in the trial will be used. The calculation of the sample size has been done with Epidat 3.1 software. Considering a significance level of 5% (Type I error), a power of 80% (complementary of the Type II error) and a minimum detectable standardized difference of means of 0.9, 30 patients per group are needed (Bonferroni correction included).

An intention-to-treat approach will be used. A descriptive analysis will be performed where quantitative variables will be described by their means and standard deviations or their medians and interquartile ranges, as appropriate. The quantitative ones will be summarized by their absolute and relative frequencies. Parametric and non-parametric tests will be employed for contrasting equality among groups.

Univariate and multivariate mixed models will be used in order to assess the effects size of the different diets (fixed effects) on the patients (random effects) unadjusted and adjusted by potential confounders, respectively. P-values under 5% will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 1 month to 2 years.
2. Children admitted to PICU.
3. Children receiving enteral nutrition with an estimated length of over 72 hours.

Exclusion Criteria: Children who met any of the following criteria will be excluded:

1. Age less than 1 month or over 2 years.
2. Diabetes mellitus or any inborn metabolic error.
3. Parenteral nutrition.
4. Bicarbonate infusion.
5. Renal replacement therapy.
6. Children receiving exclusive breastfeeding or in a need of special enteral formula.

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2016-12-28 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Nitrogen balance variation | From date of randomization until the date of first documented progression or date of discharge, whichever came first, assessed up to 7 days
  The variation of nitrogen balance (NB) from baseline to the study ending
Proportion of patients that meet study ending criteria | From date of randomization until the date of first documented progression or date of discharge, whichever came first, assessed up to 7 days
  Study ending criteria: serum urea levels elevates higher than 80 mg/dL without evidence of renal function disturbance or hypercatabolism; hyperproteinemia higher than 8.5 g/dL .

SECONDARY OUTCOMES:
variation of plasma protein levels | From date of randomization until the date of first documented progression or date of discharge, whichever came first, assessed up to 7 days
  variation of plasma protein levels (mg/dL) (total proteins, albumin, prealbumin, transferrin and retinol-binding protein)
variation of resting energy expenditure | From date of randomization until the date of first documented progression or date of discharge, whichever came first, assessed up to 7 days
  variation of resting energy expenditure measured with indirect calorimetry during the study period.
the incidence of gastrointestinal complications | From date of randomization until the date of first documented progression or date of discharge, whichever came first, assessed up to 7 days
  Gastrointestinal complications: abdominal distension, vomiting, diarrhea and excessive gastric residue

CONTACTS AND LOCATIONS:
Overall Officials: Angel P Carrillo, PhD, MD, Principal Investigator — Hospital General Universitario Gregorio Marañón. Pediatric Intensive Care Unit.
Locations (3):
- Spain (3):
  - Hospital Clínico Universitario de Santiago-CHUS, Santiago de Compostela, Galicia
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General Universitario Gregorio Marañón, Madrid

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD)
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of the study

REFERENCES:
- [Derived] Fernandez R, Urbano J, Carrillo A, Vivanco A, Solana MJ, Rey C, Lopez-Herce J. Comparison of the effect of three different protein content enteral diets on serum levels of proteins, nitrogen balance, and energy expenditure in critically ill infants: study protocol for a randomized controlled trial. Trials. 2019 Oct 11;20(1):585. doi: 10.1186/s13063-019-3686-8. PMID 31604481